CLINICAL TRIAL: NCT01009684
Title: INAS-SCORE International Active Surveillance Study - Safety of Contraceptives: Role of Estrogens
Brief Title: International Active Surveillance Study - Safety of Contraceptives: Role of Estrogens
Acronym: INAS-SCORE
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Principal Investigator, Klaas Heinemann, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2009_01
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Contraception
Keywords: Contraception; Estradiol valerate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DNG/EV: Users of the oral contraceptive containing Dienogest and Estradiol valerate
- Other OCs: Users of oral contraceptives (OCs) containing other progestins and estrogens

SUMMARY:
The primary objective of the study is to assess the risks of short and long-term use of estradiol valerate/dienogest (EV/DNG) and of established oral contraceptives (OCs) in a study population that is representative for the actual users of the individual preparations. This includes an estimate of the absolute risk of rare serious adverse outcomes.

DETAILED DESCRIPTION:
During the development of oral contraceptives (OCs) over the last decades, ethinyl-estradiol (EE) has been reduced under the hypothesis that lower EE doses lead to a better safety profile and specifically to a lower venous thromboembolism (VTE) incidence. However, the reduction of the EE dose led to a less favorable bleeding control.

Though EE has been utilized within numerous OCs, efforts have been made to utilize estradiol (E2) and estradiol valerate (EV) which have lower impact on the hepatic system and subsequently on hemostatic parameters. Bayer Schering Pharma has developed a new EV based OC in a dosing regimen that combines both reliable contraception and acceptable bleeding profile.

The INAS-SCORE study was designed as an international, prospective, controlled, non-interventional cohort study. The study was started in Europe and was extended to the US after the launch of the new regimen. New users of an OC (starters or switchers) are accrued by a network of prescribing physicians. Even in the event of high drop-out rates, a 3 to 5-year follow-up of 50,000 women should be sufficient to document about 150,000 women-years. Baseline and follow-up information are collected via a self-administered questionnaire. All self-reported clinical outcomes of interest will be validated via health care professionals. Classification of reported outcomes as "confirmed" or "unconfirmed" will be checked via blinded, independent adjudication. A multifaceted 4-level follow-up procedure proved to ensure low loss to follow-up rates.

The main clinical outcomes of interest for the short and long-term follow-up are cardiovascular events, primarily deep venous thrombosis, pulmonary embolism, acute myocardial infarction, and cerebrovascular accidents.

Data analysis will be based on life-table methods. All analyses will make allowance for confounding, using multivariate techniques such as Cox regression.

Study amendment:

Follow-up was initially expected to last until 2014 for the United States and Europe. However, the European regulatory authorities were concerned about the low proportion of Qlaira users in the United States and requested that the primary analysis should be based on the European study arm only. However, this reduction in sample size results in a reduction of the statistical power.

Therefore it was agreed upon with the European regulatory authorities to extend the follow-up period in Europe till 2016. This will ensure that the statistical power in the European study arm will be as high as the originally planned power for the complete study population (European and US study population combined). The total exposure in Europe will be sufficient to exclude a twofold risk of VTE and a threefold risk of ATE for Qlaira compared to 'Other COCs'.

ELIGIBILITY:
Inclusion Criteria:

* women who have a new prescription for an OC
* women who are willing to participate in this long-term follow-up study

Exclusion Criteria:

* women who are not cooperative
* women with a language barrier

There are no specific medical inclusion or exclusion criteria.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants are recruited by their attending gynecologists. The sample should be representative of users of oral contraceptives (OCs).
Sampling Method: Non-Probability Sample
Enrollment: 50203 (Actual)
Dates: Start 2009-08; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Venous Thromboembolic Events (VTE) | up to 7 years
Acute Myocardial Infarction (AMI) | up to 7 years
Cerebrovascular Accidents (CVA) | up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, PhD, MD, MSc, Principal Investigator — Berlin Center for Epidemiology and Health Research
Locations (1):
- Berlin Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Result] Dinger J, Do Minh T, Heinemann K. Impact of estrogen type on cardiovascular safety of combined oral contraceptives. Contraception. 2016 Oct;94(4):328-39. doi: 10.1016/j.contraception.2016.06.010. Epub 2016 Jun 22. PMID 27343748
- [Result] Barnett C, Hagemann C, Dinger J, Do Minh T, Heinemann K. Fertility and combined oral contraceptives - unintended pregnancies and planned pregnancies following oral contraceptive use - results from the INAS-SCORE study. Eur J Contracept Reprod Health Care. 2017 Feb;22(1):17-23. doi: 10.1080/13625187.2016.1241991. Epub 2016 Oct 17. PMID 27749101